CLINICAL TRIAL: NCT03605472
Title: Comparison of Cervical Ultrasound and Echoscintigraphy for Preoperative Localization Diagnosis in Primary Hyperparathyroidism
Acronym: ECHOPARAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA17094
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Primary Hyperparathyroidism
Keywords: primary hyperparathyroidism; cervical ultrasound; echoscintigraphy
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: cervical ultrasound

INTERVENTIONS:
Other: cervical ultrasound — cervical ultrasound will be realized by a endocinologist trained in the cervical ultrasound

SUMMARY:
The biological diagnosis of the primary hyperparathyroidism is now facilitated by the reliability of the balance of phosphate and calcium and the dosage of parathyroid hormone (PTH).

This diagnosis of preoperative localization is important as surgery are now targeted to the responsible lesion.

The "gold standard" for this localization is the cervical ultrasound exploring the usual sites of adenomas and a MIBI scintigraphy (the parathyroid adenoma significantly concentrating this cell marker).

However, the diagnosis of preoperative localization remains a subject of discussion as to the most appropriate tests. Indeed, the morphological diagnosis is performed at the ultrasound stage in more than half the cases. It is the new performance of this morphological examination that makes it possible to obtain these results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hyperparathyroidism with surgery indication
* Age > 18yo

Exclusion Criteria:

* surgical contraindication
* medical treatment by cinacalcet
* non sporadic hyperparathyroidism
* Age <18yo
* Protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-10-05 (Estimated); Study Completion 2020-03-05 (Estimated)

PRIMARY OUTCOMES:
Adenoma parathyroid diagnosed using cervical ultrasound | Day 0
  Adenoma parathyroid diagnosed using cervical ultrasound. Cervical ultrasound will be realized by a endocrinologist trained in the cervical ultrasound and not informed of the results of the echoscintigraphy
Adenoma parathyroid diagnosed using echoscintigraphy | Day 0
  Adenoma parathyroid diagnosed using echoscintigraphy. Echoscintigraphy will be realized by a nuclear physician not informed of the results of the cervical ultrasound
Adenoma parathyroid diagnosed using anatomopathology | Day 0
  Adenoma parathyroid diagnosed by anatomopathologist, after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France